CLINICAL TRIAL: NCT02775539
Title: Beta3 Adrenergic Agonist Treatment in Chronic Pulmonary Hypertension Secondary to Heart Failure
Brief Title: Beta3 Agonist Treatment in Chronic Pulmonary Hypertension Secondary to Heart Failure
Acronym: SPHERE-HF
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fundación Centro Nacional de Investigaciones Cardiovasculares Carlos III (Other)
Collaborators: Hospital Clinic of Barcelona (Other); Hospital Universitario 12 de Octubre (Other); Puerta de Hierro University Hospital (Other); Fundació Institut de Recerca de l'Hospital de la Santa Creu i Sant Pau (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: SPHERE-HF
Record Dates: First submitted 2016-05-14; First posted 2016-05-17 (Estimated); Last update posted 2016-05-17 (Estimated); Status verified 2016-05

CONDITIONS: Pulmonary Hypertension; Mirabegron; Heart Failure; Pulmonary Vascular Resistance Abnormality
Keywords: Pulmonary hypertension; Mirabegron; Heart failure; B3 adrenergic
MeSH Terms: conditions — Hypertension, Pulmonary; Heart Failure | interventions — mirabegron

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Mirabegron (Active Comparator): Oral mirabegron, starting with 50 mg once a day and titrated till a maximum of 200 mg once a day.
  Interventions: Drug: Mirabegron
- Placebo (Placebo Comparator): Oral placebo, similarly titrated to ensure blindness.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Mirabegron — Patients will receive 50 to 200 mg of mirabegron once a day during 16 weeks. Dose will be titrated during the first 8 weeks.
  Arms: Mirabegron
Drug: Placebo
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of mirabegron (a B3 adrenergic receptor agonist) in patients with pulmonary hypertension secondary to heart failure by conducting a randomized multicenter phase II placebo-controlled clinical trial.

DETAILED DESCRIPTION:
Pulmonary hypertension (PH) affects 60-80% of patients with chronic heart failure (HF) and has a critical impact on prognosis. Currently, there is no specific treatment approved for this indication. Experimental research, performed by members of the consortium, demonstrates that treatment with B3 adrenergic receptor agonists produces a beneficial effect on pulmonary hemodynamics, right ventricular (RV) remodeling and pulmonary vascular proliferation in a translational pig model of postcapillary PH. Mirabegron, an oral B3AR agonist, is currently approved for a different medical condition (overactive bladder syndrome) with a good safety profile. Our main objective is to evaluate the efficacy and safety of mirabegron in patients with PH secondary to HF.

The objective will be evaluated by conducting a phase-2 randomized placebo-controlled clinical trial in patients with PH associated to HF. Patients will be randomized 1:1 to mirabegron or placebo, and dose will be titrated till 200 mg/day. Patients will be evaluated with quality of life questionnaire, blood analysis, ECG, echocardiography, 6-minute walking test, right heart catheterization (RHC) and cardiac magnetic resonance (CMR) at baseline and after 16 weeks of treatment.

ELIGIBILITY:
Inclusion Criteria:

* Written inform consent;
* >18 years-old;
* HF with reduced or preserved ejection fraction, according to the definition of the European Society of Cardiology guidelines.
* Severe PH and/or combined postcapillary and precapillary PH (also knows as reactive or out-of-proportion PH) determined by RHC showing the following:

  * Pulmonary arterial wedge pressure or end-diastolic left ventricular pressures ≥15 mmHg;
  * Mean PAP≥25, and:
  * PVR≥3 UW and/or diastolic gradient≥7 mmHg or
  * Transpulmonary gradient≥12.
* NYHA functional class II-IV;
* On optimized evidence-based pharmacological treatment;
* Stable clinical condition defined as no changes in therapeutic regimen or hospitalization in the 30 days preceding recruitment and no current plan for changing therapy.

Exclusion Criteria:

* Non-coronary cardiac surgery or non-coronary percutaneous procedure within the 12 months preceding recruitment or programmed;
* Myocardial infarction or coronary revascularization during the last 3 months,
* Myocardial resynchronization therapy initiated during the last 6 months;
* Sinus tachycardia or atrial fibrillation with uncontrolled heart rate (>100 bpm);
* Uncontrolled hypertension (PAS>180 or PAD>110 mmHg) or symptomatic hypotension (PAS<90 mmHg).
* Infiltrative myocardial disease.
* Expected survival <1 year due to a disease other than PH;
* Severe renal failure (GFR <30 mL/min/1.73 m2 or haemodialysis);
* Severe hepatic impairment (serum aspartate aminotransferase (AST) and/or alanine aminotransferase (ALT) >3x the upper limit of normality at screening;
* cQT interval on the ECG >430 ms in male or >450 ms in female;
* Concomitant use of specific pulmonary vasodilator therapy (i.e. endothelin receptor antagonists, phosphodiesterase -5 inhibitors, guanylate cyclase stimulators).
* Concomitant use of digoxin, flecainide, propafenone, dabigatran, tricycle antidepressants, or another strong inhibitors of CYP2D6 (with the exception of betablockers).
* Significant obstructive lung disease (FEV1/FVC<0.7 associated with FEV1<50% of predicted value).
* Significant restrictive lung disease (TLC<60%).
* Participation in another clinical trial.
* Female with childbearing potential.
* Known hypersensitivity to mirabegron or to any of its excipients.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2016-06; Primary Completion 2017-01 (Estimated); Study Completion 2019-06 (Estimated)

PRIMARY OUTCOMES:
Change in pulmonary vascular resistance (PVR) from baseline to week 16 assessed by right heart catheterization (RHC). | 16 weeks

SECONDARY OUTCOMES:
Change from baseline in 6-minute walking distance | 16 weeks
Change from baseline in NYHA functional class | 16 weeks
Change from baseline in quality of life | 16 weeks
Change from baseline in dyspnea Borg score | 16 weeks
Change from baseline in mean PAP as assessed by RHC | 16 weeks
Change from baseline in cardiac index (CI) as assessed by RHC and cardiac magnetic resonance (CMR) | 16 weeks
Change from baseline in RV ejection fraction as assessed by CMR | 16 weeks
Change from baseline in BNP/NT-proBNP | 16 weeks
Hospital admissions due to worsening cardiopulmonary status | 16 weeks
Mortality | 16 weeks
Urgent heart transplantation | 16 weeks
New onset arrhythmia | 16 weeks
Need for initiation of intravenous therapy due to worsening HF | 16 weeks
Adverse drug effects | 16 weeks

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Garcia-Lunar I, Blanco I, Fernandez-Friera L, Prat-Gonzalez S, Jorda P, Sanchez J, Pereda D, Pujadas S, Rivas M, Sole-Gonzalez E, Vazquez J, Blazquez Z, Garcia-Picart J, Caravaca P, Escalera N, Garcia-Pavia P, Delgado J, Segovia-Cubero J, Fuster V, Roig E, Barbera JA, Ibanez B, Garcia-Alvarez A. Design of the beta3-Adrenergic Agonist Treatment in Chronic Pulmonary Hypertension Secondary to Heart Failure Trial. JACC Basic Transl Sci. 2020 Mar 11;5(4):317-327. doi: 10.1016/j.jacbts.2020.01.009. eCollection 2020 Apr. PMID 32368692